CLINICAL TRIAL: NCT01828190
Title: Prospective Open-label Study of the Efficacy of the Addition of Hyperbaric Oxygen to the Treatment of Patients With Perianal Fistulas Already Treated With TNF Alpha Blockers
Brief Title: The Influence of Hyperbaric Oxygen in Patients With Perianal Crohn's Disease Already Treated With TNF Alpha Blockers Treated With TNF Alpha Blockers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HBOT- fistulas non-naive
Record Dates: First submitted 2013-04-08; First posted 2013-04-10 (Estimated); Last update posted 2023-03-22 (Actual); Status verified 2013-04

CONDITIONS: Crohn's Disease; Perianal Fistulas
Keywords: crohn's disease; perianal fistulas; TNF alpha blockers; hyperbaric oxygen therapy
MeSH Terms: conditions — Crohn Disease | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hyperbaric oxygen (Experimental): hyperbaric oxygen therapy will be given for 2 months. TNF alpha blocker therapy will remain the treatment received before recruitment.
  Interventions: Other: Hyperbaric oxygen

INTERVENTIONS:
Other: Hyperbaric oxygen — HBOT will be given for 40 sessions of 2 atmospheres for 90 minutes each session, 5 times a week (2 months). TNF alpha blocker therapy will remain the treatment received before recruitment.

SUMMARY:
The aim of this study is to evaluate the effect of hyperbaric oxygen therapy (HBOT) on patient suffering from residual Crohn's disease related perianal fistulas already treated with TNF alpha blockers

DETAILED DESCRIPTION:
This study is a prospective open-label study that consists three periods: screening, treatment and follow-up. After signing an informed consent, subjects will be assessed by a gastroenterologist, a surgeon (for the diagnosing the perianal disease and assessing the need for surgery) and a HBOT specialist for assessing the capability of the subject to undergo HBOT treatment.After the screening period, eligible subjects will enter an 8 weeks HBOT treatment period, combined with TNFalpha blocker treatment. This period will be followed by a 4 months follow-up period in which treatment with TNFalpha blocker will continue.

All patients will have an MRI and TRUS examinations to assess the fistulas and also blood tests for CBC, chemistry, inflammatory markers and cytokine analysis. Same evaluation will be repeated at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

patients aged 18 and above that suffer from Crohn's disease one or more perianal draining fistulas for at least 3 months currently receiving a TNFalpha blocker for at least 3 months (without improvement of the perianal disease)

Exclusion Criteria:

Pregnancy or plans to conceive during the next year Inability (such as previous adverse effects, tuberculosis, concurrent infection etc.)or unwillingness to start or continue with TNF alpha blockers treatment.

Any past or current malignancy Treatment with HBOT in the last year Claustrophobia Middle ear problems Inability to equalize pressure in the middle ear Medical status that precludes treatment with HBOT such as chest X-ray abnormality, epilepsy, severe congestive heart failure, uncontrolled diabetes or uncontrolled hypertension Any perianal surgery in the last 6 months Any change in Crohn's disease medications in the last 3 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-03; Primary Completion 2015-03 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Reduction of fistulas number | 0, 32 weeks
  As assessed by MRI and TRUS

SECONDARY OUTCOMES:
Reduction of perianal symptoms | 0, 4, 8, 14, 20, 32
  As assessed by PDAI score

CONTACTS AND LOCATIONS:
Overall Officials: Haim Shirin, MD, Principal Investigator — Assaf Harofe Medical Center
Locations (1):
- The institute of gastroenterology and liver disease, Assaf Harofe Medical Center, Ẕerifin, Israel